CLINICAL TRIAL: NCT00813124
Title: Azacitidine Maintenance Therapy After Allogeneic Stem Cell Transplantation for Chronic Myelogenous Leukemia (CML)
Brief Title: Azacitidine After Allo Blood And Marrow Transplantation (BMT) for Chronic Myelogenous Leukemia (CML)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-0087; NCI-2012-02122 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2008-12-18; First posted 2008-12-22 (Estimated); Results first posted 2021-01-07 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-01

CONDITIONS: Stem Cell Transplantation; Leukemia
Keywords: Chronic Myelogenous Leukemia; CML; Donor stem cell transplant; Allogeneic stem cell transplantation; Stem cell transplant; ATG; Antithymocyte globulin; Vidaza; Azacitidine; 5-Azacitidine; 5-Aza; 5-AZC; Ladakamycin; NSC-102816; allotx; Busulfan; Busulfex; Myleran; Fludarabine; Fludarabine Phosphate; Tacrolimus; Methotrexate; Azacitidine maintenance therapy; molecular remission; HLA compatible donor; Engraftment; Chimerism; Graft vs host disease; GVHD
MeSH Terms: conditions — Leukemia; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Graft vs Host Disease | interventions — fludarabine; fludarabine phosphate; Busulfan; thymoglobulin; Antilymphocyte Serum; Azacitidine; Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Azacytidine Maintenance after allotx (Experimental): Busulfan + Fludarabine + ATG + Azacytidine after allogeneic stem cell transplantation (allotx)
  Interventions: Drug: Fludarabine; Drug: Busulfan; Drug: Thymoglobulin; Drug: Azacitidine; Procedure: Stem Cell Transplant

INTERVENTIONS:
Drug: Fludarabine — 40 mg/m^2 by vein over 60 minutes on Day -5 through Day -2.
  Other Names: Fludarabine Phosphate
Drug: Busulfan — Busulfan administered at the dose calculated to achieve an area under curve (AUC) of 4000 µMol-min + 12% based on the pharmacokinetic studies (days -5, -4, -3, and -2).
  Other Names: Busulfex; Myleran
Drug: Thymoglobulin — 2.5 mg/kg by vein over about 4-6 hours on Day -3 through Day -1.
  Other Names: Antithymocyte globulin; ATG
Drug: Azacitidine — Start cycles of 32 mg/m^2 daily as an injection under the skin once a day over 5 days in a row, starting about 5 weeks after the transplant. This may be repeated once a month for up to 4 months after the transplant.
  Other Names: 5-Azacitidine; 5-Aza; 5-AZC; Ladakamycin; NSC-102816; Vidaza
Procedure: Stem Cell Transplant — Stem cell infusion on day 0 administered by vein after collected from donor.
  Other Names: allotx; allogeneic stem cell transplantation

SUMMARY:
The goal of this clinical research study is to learn if Vidaza (azacitidine) when given to patients with CML after an donor stem cell transplant will increase the likelihood of achieving a complete remission of CML.

DETAILED DESCRIPTION:
Study Drug:

Azacitidine is designed to block genes in cancer cells that stop the function of the tumor-fighting genes. By blocking the "bad" genes, the tumor-fighting genes may be able to work better.

Study Drug Administration and Procedures before the Stem Cell Transplant:

If you are found to be eligible to take part in this study, you will be given chemotherapy before the transplant of donor cells. The chemotherapy is designed to kill leukemia cells and will also block your body's ability to reject the donor cells that will be given to you during the transplant. You will receive the chemotherapy on the days before the transplant. You will receive the transplant on Day 0.

This low-level test dose of busulfan is to check how fast busulfan is processed by your body and cleared from your blood. This information will help the doctor decide the dose of busulfan you will receive. You may receive the busulfan test dose as an outpatient during the week before you are admitted to the hospital or as an inpatient on Day -8 (8 days before your stem cell transplant).

About 11 samples of blood (about 1 teaspoon each time) will be drawn for pharmacokinetic (PK) testing. PK testing measures the amount of study drug in the body at different time points. These blood samples will be drawn at various times before you receive busulfan and over the next 11 hours. These blood draws will be repeated again on the first day of high-dose busulfan treatment (Day -5).

A heparin lock line (small IV line) will be placed in your vein to lower the number of needle sticks needed for these draws. If it is not possible for the PK tests to be performed for technical or scheduling reasons, you will receive the standard fixed dose of busulfan.

On Days -5 through -2, you will receive fludarabine by vein over 1 hour, then busulfan by vein over 3 hours.

If you are going to be receiving a transplant from an unrelated donor, or if you have a donor that is mismatched, you will also receive antithymocyte globulin (ATG) by vein over 4 hours on the 3 days before the transplant. This drug is designed to further weaken your immune system to reduce the risk of rejecting of the transplant.

Stem Cell Transplant:

After the blood-forming cells are collected from the donor, they will be given to you by vein. You will be given standard drugs to help decrease the risk of side effects. You may ask the study staff for information about how the drugs are given and their risks.

Drugs to Prevent Infections:

You will receive several drugs to help the stem cell transplant work and to help decrease the risks of infections while your immune system is weak. Tacrolimus and methotrexate will be given to decrease the risk of graft-versus-host disease (GVHD), a problem that may occur if the donor's immune cells fight your body.

* Tacrolimus will be started 2 days before the transplant and will continue for as long as your doctor thinks is necessary. This is usually 3-12 months, but may be longer if you develop GVHD. Tacrolimus is given by vein non-stop until you are able to eat. Once you can eat, it will be given by mouth.
* Methotrexate is given by vein over about 15-30 minutes on Days 1, 3, 6, and 11.

Several drugs will also be given to decrease the risk of other infections. Some of these antibiotics are given by vein, and some are given as pills. The length of time that you will take the antibiotics will vary. Your doctor will describe this to you in more detail.

Study Drug Administration after the Stem Cell Transplant:

You will receive azacitidine as an injection under the skin once a day over 5 days in a row, starting about 5 weeks after the transplant. This may be repeated once a month for up to 4 months after the transplant. You will have about 23 days of "rest" between each cycle of treatment (a cycle is the period of 28 days). If intolerable side effects occur, treatment with azacitidine may be interrupted or stopped altogether.

Study Visits:

You will be in the hospital for about 3-4 weeks after the transplant. You will have check-ups every day until you leave the hospital. After you leave, the number of study visits will vary, depending on your condition.

You will have bone marrow aspirations collected before chemotherapy, around 1, 6, and 12 months after the transplant. To collect a bone marrow aspirate, an area of the hip bone is numbed with anesthetic, and a small amount of bone marrow is withdrawn through a large needle. The bone marrow samples will be used to check the status of the disease and to learn the way azacitidine works.

Blood (about 2 teaspoons each time) will be drawn to learn about patterns of a process called methylation. Methylation is a process by which the body may turn "on and off" certain genes. Blood will be drawn at the following times:

* At baseline.
* Before the stem cell transplant (Day 0).
* Six (6), 9, and 12 months after the transplant.
* Before you receive your first dose of azacitidine (Day 1 of each cycle).
* After you receive the last dose of azacitidine (Day 5 of each cycle).

Blood (about 8 teaspoons each time) will be drawn to learn about the body's immune system recovery, at the following times:

* Cycle 1- Day 1
* Cycle 1 - Day 14
* Cycle 3 - Day 1

Length of Study:

You will remain on study for up to 1 year. You may be taken off study early if the disease gets worse or intolerable side effects occur.

This is an investigational study. Azacitidine is FDA approved and commercially available in patients with myelodysplastic syndrome. Its use in patients with CML is investigational. All other drugs used in this study are FDA approved and commercially available.

Up to 57 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with age <= 75 years with CML in first chronic phase, which has failed to achieve a cytogenetic or molecular complete remission or has progressed after imatinib treatment. Criteria for failure are the international consensus criteria (Appendix H). Patients intolerant to tyrosine kinase inhibitor therapy are also eligible.
2. Patients with age <= 75 with CML in accelerated phase or blast crisis that have <= 15% blasts in the blood and bone marrow at study entry.
3. Donor: HLA-compatible related (HLA-A, -B, -DRB1 matched or with one-antigen mismatch) or HLA-compatible unrelated (HLA-A, -B, -C and -DRB1 matched or with one-antigen mismatch).
4. Age 18 to 75 years.
5. Zubrod performance status <= 2.
6. Left ventricular ejection fraction => 40%.
7. Pulmonary function test within the following parameters: forced expiratory volume at one second (FEV1), forced vital capacity (FVC) and diffusing capacity of lung for carbon monoxide (DLCO) => 50% of expected, corrected for hemoglobin.
8. Serum creatinine < 1.5 mg/dL or creatinine clearance greater or equal than 40 cc/min.
9. Serum direct bilirubin < 1.5 mg/dL (unless Gilbert's syndrome)
10. Serum glutamate pyruvate transaminase (SGPT) <= 200 IU/L unless related to patient's malignancy.
11. Patients treated with any tyrosine kinase inhibitor, interferon or any experimental therapy are eligible.
12. Patients with age <75 years with CML in second or subsequent chronic phase.

Exclusion Criteria:

1. Uncontrolled infection, not responding to appropriate antimicrobial agents after seven days of therapy.
2. Pleural/pericardial effusion or ascites estimated to be >1L.
3. HIV-positive.
4. Breast feeding or pregnancy. Pregnancy means a positive beta human chorionic gonadotropin (HCG) test in a woman with child bearing potential defined as not post-menopausal for 12 months or no previous surgical sterilization.
5. Known or suspected hypersensitivity to azacitidine or mannitol.
6. Patients with advanced malignant hepatic tumors.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-12; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard E. Champlin, MD, BS, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: December 17, 2008 to February 27, 2014. All recruitment done at The University of Texas (UT) MD Anderson Cancer Center.
Groups:
- Azacitidine Post Transplant: Fludarabine 40 mg/m^2 intravenous (IV) Day -5 to Day -2; Busulfan dose calculated to achieve area under curve (AUC) of 4000 µMol-min + 12% based on pharmacokinetic studies (days -5, -4, -3, and -2); Thymoglobulin: 2.5 mg/kg IV on Day -3 to Day -1; Azacitidine 32 mg/m^2 subcutaneous daily for 5 days starting 5 weeks after transplant, repeated monthly up to 4 months. Allogeneic stem cell infusion (allotx) on day 0.
Period: Overall Study
Arm/Group | Azacitidine Post Transplant
Started | 24
Completed | 12
Not Completed | 12
Not completed — Death | 2
Not completed — Ineligible - Participants did not received Azacytidine | 9
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Azacytidine Maintenance After Allotx: Fludarabine 40 mg/m^2 intravenous (IV) Day -5 to Day -2; Busulfan dose calculated to achieve area under curve (AUC) of 4000 µMol-min + 12% based on pharmacokinetic studies (days -5, -4, -3, and -2); Thymoglobulin: 2.5 mg/kg IV on Day -3 to Day -1; Azacitidine 32 mg/m^2 subcutaneous daily for 5 days starting 5 weeks after transplant, repeated monthly up to 4 months. Allogeneic stem cell infusion (allotx) on day 0.
Arm/Group | Azacytidine Maintenance After Allotx
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Molecular Response
Description: Molecular Remission defined as two consecutive bone marrow samples done one month apart with negative PCR( polymerase chain reaction) tor CML.
Time Frame: 12 month post BMT
Measure: Count of Participants; unit: Participants
Arm/Group | Azacytidine Maintenance After Allotx
Number analyzed (Participants) | 12
Participants
  Complete Response | 8
  Partial Response | 0
  Progressive Disease | 4

ADVERSE EVENTS:
Time Frame: Adverse event data collected through four treatment cycles of 28 days.
Arm/Group | Azacytidine Maintenance After Allotx
All-Cause Mortality (participants affected / at risk) | 2/24
Serious Adverse Events (participants affected / at risk) | 14/24
Other Adverse Events (participants affected / at risk) | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Azacytidine Maintenance After Allotx (N=24)
ALT increased (Investigations) | 2
Bacterial (Infections and infestations) | 6
Confusion (Psychiatric disorders) | 1
Delayed engraftment (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Fungal (Infections and infestations) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2
Hemorrhagic Cystitis (Renal and urinary disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Low granulocyte (Blood and lymphatic system disorders) | 1
Low platelet (Investigations) | 2
Rash (Skin and subcutaneous tissue disorders) | 2
Thromboembolic event (Vascular disorders) | 2
Viral (Infections and infestations) | 5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Azacytidine Maintenance After Allotx (N=24)
Abdominal pain (Gastrointestinal disorders) | 2
ALT increased (Investigations) | 7
Anorexia (Metabolism and nutrition disorders) | 1
Bacterial (Infections and infestations) | 4
Blurred vision (Eye disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 3
Broncholitis obliterans (Respiratory, thoracic and mediastinal disorders) | 1
Bruising (Injury, poisoning and procedural complications) | 1
Creatinine increased (Investigations) | 3
Diarrhea (Gastrointestinal disorders) | 7
Dizziness (Nervous system disorders) | 1
Dry eye (Eye disorders) | 2
Fever (General disorders) | 18
Flu like syndrome (General disorders) | 1
Fluid overload (General disorders) | 5
Headache (Nervous system disorders) | 5
Hemorrhagic Cystitis (Renal and urinary disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypertension (Vascular disorders) | 2
Low granulocyte (Blood and lymphatic system disorders) | 1
Low platelet (Investigations) | 2
Nausea (Gastrointestinal disorders) | 22
Oral mucositis (Gastrointestinal disorders) | 14
Rash (Skin and subcutaneous tissue disorders) | 10
T bilirubin increased (Investigations) | 5
Viral (Infections and infestations) | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes